CLINICAL TRIAL: NCT06052176
Title: Randomized Clinical Trial in Hepatic Encephalopathy to Study Lasting Cognitive Improvement With Intravenous Albumin
Brief Title: Hepatic Encephalopathy and Albumin Lasting Cognitive Improvement
Acronym: HEAL-LAST
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Hunter Holmes Mcguire Veteran Affairs Medical Center (U.S. Federal Agency)
Collaborators: Grifols Biologicals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: Double | Purpose: Prevention
Other Study IDs: BAJAJ0035
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis; Hepatic Encephalopathy
Keywords: albumin; cirrhosis; inflammation; cognitive performance
MeSH Terms: conditions — Fibrosis; Hepatic Encephalopathy; Inflammation | interventions — Albumins

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Subjects will be blinded to which infusions are albumin versus placebo. All infusion tubing and bag will be covered in foil and the subjects will not be aware of the timing of the saline vs albumin infusion to maintain blinding for the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Saline given at the same volume as the albumin on visits the patients are assigned to it
  Interventions: Drug: Albumin Infusion
- Albumin (Active Comparator): IV Albumin at 1.5g/kg ideal body weight
  Interventions: Drug: Albumin Infusion

INTERVENTIONS:
Drug: Albumin Infusion — Intravenous human serum albumin to be given at 1.5g/kg ideal body weight
  Other Names: Albutein

SUMMARY:
Hypothesis: Improvement in cognitive dysfunction with IV albumin in patients with cirrhosis with prior HE and MHE lasts for several weeks after albumin infusion has ended, and is due to persistent improvement in inflammatory markers, endothelial dysfunction, albumin function and gut microbial changes.

This will be a single-arm, single-blind sequential trial of IV 25% albumin and IV saline over 8 weeks with biological sampling and cognitive and health related quality of life (HRQOL) testing with each subject acting as their own control.

DETAILED DESCRIPTION:
In outpatients with cirrhosis with prior HE who have cognitive impairment despite adequate therapy, how long the impact of albumin lasts and through which potential mechanism(s) needs to be determined.

A prior recent HEAL trial showed that patients with prior HE and current minimal hepatic encephalopathy (MHE) randomized to albumin experienced significant improvement in cognitive dysfunction and psychosocial quality of life. Moreover, these improvements persisted a week after the last albumin infusion, which was not seen in the placebo group. This was accompanied by an improvement in endothelial dysfunction, ischemia-modified albumin levels and inflammatory markers that persisted one week even after albumin discontinuation. The reported half-life of IV albumin is 2 weeks, but the function and the length of time of albumin's action in decompensated cirrhosis is lower, and further details surrounding albumin pharmacokinetics in this population remain unelucidated. The mechanisms and length of time albumin's potential improvement for patients with MHE after treatment discontinuation also require continued study.

Study design:

This will be a single-arm, single-blind sequential trial of IV 25% albumin and IV saline over 8 weeks with biological sampling and cognitive and health related quality of life (HRQOL) testing with each subject acting as their own control.

Th order of the albumin and placebo infusion and blind the infusions from the subjects and the assessors of the outcomes will be changed.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Cirrhosis diagnosed using either (a) liver biopsy, (b) transient wave elastography (>20 KPa) (c) radiological evidence consistent with cirrhosis, (d) in a patient with chronic liver disease endoscopic or radiological evidence of varices (e), in a patient with chronic liver disease, platelet count <150,000/mm3 and AST/ALT ratio >1.
* Cognitive impairment defined by MHE on psychometric hepatic encephalopathy score (PHES), critical flicker frequency (CFF), or EncephalApp Stroop
* Prior HE controlled by lactulose or rifaximin for at least one month
* Serum albumin <4gm/dl

Exclusion Criteria:

* Unclear diagnosis of cirrhosis
* No prior overt HE
* No cognitive impairment on the tests noted
* Requiring regular albumin infusions within 3 months or anticipated during the study visit
* Infection within a month
* Allergies to albumin
* Unlikely to be adherent to the study
* Unable or unwilling to consent
* West Haven Criteria>2
* Alcohol abuse within 1 month
* Serum albumin >4gm/dl
* Congestive heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Delta change in Psychometric Hepatic Encephalopathy Score (PHES) in Placebo phase vs Albumin phase | 4 weeks each
  cognitive improvement (PHES score ranges from -15 to 5), higher is good

SECONDARY OUTCOMES:
EncephalApp Stroop change in Placebo phase vs Albumin phase | 4 weeks each
  cognitive improvement (Stroop OffTime+OnTime in seconds will be evaluated); higher is worse
Critical Flicker Frequency change in Placebo phase vs Albumin phase | 4 weeks each
  cognitive improvement (Hz at which CFF is reached will be evaluated), higher is good
Change in Sickness Impact Profile Placebo phase vs Albumin phase | 4 weeks each
  Health-related quality of life change (SIP total, psychosocial and physical scores where a higher score indicates poor HRQOL willl be evaluated)
Change in PROMIS-29 Placebo phase vs Albumin phase | 4 weeks each
  Health-related quality of life change (Total PROMIS-29 score will be evaluated)
Change in MELD-Na score Placebo phase vs Albumin phase | 4 weeks each
  Liver disease severity change using MELD-Na; higher is worse
Change in endotoxin binding protein Placebo phase vs Albumin phase | 4 weeks each
  Change in endotoxin binding protein will be recorded in the serum; higher is worse
Change in oxidized albumin Placebo phase vs Albumin phase | 4 weeks each
  Change in oxidized albumin will be recorded in the serum ; higher is worse
Change in ischemia modified albumin Placebo phase vs Albumin phase | 4 weeks each
  Change in ischemia modified albumin will be recorded in the serum
Change in stool bile acids Placebo phase vs Albumin phase | 4 weeks each
  Change in stool bile acids (total, primary, secondary, conjugated/deconjugated) will be recorded
Change in serum bile acids Placebo phase vs Albumin phase | 4 weeks each
  Change in serum bile acids (total, primary, secondary, conjugated/deconjugated) will be recorded
Change in serum Short-chain fatty acids Placebo phase vs Albumin phase | 4 weeks each
  Change in serum Short-chain fatty acids (acetate, propionate, butyrate will be recorded
Change in stool Short-chain fatty acids Placebo phase vs Albumin phase | 4 weeks each
  Change in stool Short-chain fatty acids (acetate, propionate, butyrate will be recorded
Change in stool bacterial alpha diversity Placebo phase vs Albumin phase | 4 weeks each
  Change in Shannon diversity of stool bacteria
Change in serum inflammatory cytokines Placebo phase vs Albumin phase | 4 weeks each
  Change in IL-6, TNF-α, IL-10, IL-1β in serum

CONTACTS AND LOCATIONS:
Locations (1):
- Hunter Holmes McGuire VA Medical Center, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No